CLINICAL TRIAL: NCT03644485
Title: Clinical Outcome of Delayed or Standard Prograf Together With Induction Therapy Followed by Conversion to Advagraf in Donation After Cardiac (or Circulatory) Death (DCD) Kidney Transplant Recipients: A Randomized, Open-label, Multicenter Clinical Trial
Brief Title: Clinical Outcome of Delayed or Standard Prograf Together With Induction Therapy Followed by Conversion to Advagraf in Donation After Cardiac (or Circulatory) Death (DCD) Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 506-MA-3186
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplant
Keywords: kidney transplant; Tacrolimus; Prograf; Advagraf; FK506
MeSH Terms: interventions — Tacrolimus; Neoadjuvant Therapy; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Prograf group (Experimental): Participants received from day 1 tacrolimus immediate-release formulation (Prograf) 0.1 - 0.15 milligrams/kilograms/day (mg/kg/day) orally at 12-hour interval (twice daily 1 hour before meal or 2 hours after meal) for approximately 1 month. At 1 month after Kidney transplant, Prograf was converted to Advagraf on a 1:1 (mg: mg) total daily dose basis. The Advagraf was administered orally once daily in the morning, 1 hour before the breakfast; the whole blood target trough level for Advagraf was maintained as 6 - 12 nanograms/milliliter(ng/mL) within months 2 to 3, and 6 - 8 ng/mL within months 4 to 6.
  Interventions: Drug: Tacrolimus immediate-release formulation; Drug: Tacrolimus prolonged-release formulation; Drug: Induction therapy; Drug: Mycophenolic acid drugs; Drug: Corticosteroids
- Delayed Prograf group (Experimental): Participants received from day 3 to 5 Prograf 0.1 - 0.15 mg/kg/day orally at 12-hour interval (twice daily 1 hour before meal or 2 hours after meal) for approximately 1 month. At 1 month after Kidney transplant, Prograf was converted to Advagraf on a 1:1 (mg: mg) total daily dose basis. The Advagraf was administered orally once daily in the morning, 1 hour before the breakfast; the whole blood target trough level for Advagraf was maintained as 6 - 12 ng/mL within months 2 to 3, and 6 - 8 ng/mL within months 4 to 6.
  Interventions: Drug: Tacrolimus immediate-release formulation; Drug: Tacrolimus prolonged-release formulation; Drug: Induction therapy; Drug: Mycophenolic acid drugs; Drug: Corticosteroids

INTERVENTIONS:
Drug: Tacrolimus immediate-release formulation — oral
  Other Names: Prograf; FK506
Drug: Tacrolimus prolonged-release formulation — oral
  Other Names: Advagraf; FK506
Drug: Induction therapy — All participants will receive induction therapy. The dosage and administration of induction immunotherapy will be a single kind of drug determined by the investigator.
Drug: Mycophenolic acid drugs — All participants will receive mycophenolic acid drugs in combination with corticosteroids. The dosage and administration of mycophenolic acid will be determined by the investigator.
Drug: Corticosteroids — All participants will receive corticosteroids in combination with mycophenolic acid drugs. The dosage and administration of corticosteroids will be determined by the investigator.

SUMMARY:
The purpose of this study is to confirm non-inferiority of delayed Prograf treatment to standard Prograf treatment in the incidence of delayed graft function (DGF) within 1 week between the 2 immunosuppressive (IS) treatment groups: delayed or standard Prograf together with induction therapy, and then convert to Advagraf usage in donation after cardiac (or circulatory) death (DCD) kidney transplant recipients.

This study will also compare the clinical outcome within 6 month post-transplant between the 2 IS treatment groups and compare the safety throughout study period between the 2 IS treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject has end-stage kidney disease who is a suitable candidate for primary DCD kidney transplantation.
* Subject is a resident of China.
* Subject is scheduled to undergo DCD renal allograft transplantation with compatible ABO blood type.
* Subject has peak panel-reactive antibodies (PRA) < 10% or "Negative" test result.
* Subject must be a recipient of a DCD kidney and receive the organ distributed by China Organ Transplant Response System only.
* Female subject must either:

  * Be of non-childbearing potential: Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or documented surgically sterile
  * Or, if of childbearing potential: Agree not to try to become pregnant throughout the study period and have a negative blood pregnancy test at screening.
* A sexually active male or female subject is utilizing highly effective forms of birth control starting at screening and throughout the study period if the risk of conception exists.
* Subject agrees not to participate in another interventional study while participating in the present study from 1 month before randomization to 1 month after the last dose of investigational drug.

Exclusion Criteria:

* Subject has previously received or is receiving an organ transplant other than kidney.
* Subject is receiving double-kidney transplant.
* Recipients of Maastricht Class I, II, and V donor organs.
* Recipients of Maastricht Class III and IV donor organs without a full complement of intensive care unit and intraoperative records.
* Subject has cold ischemia time of allograft > 24 hours before kidney transplantation surgery.
* Subject has known contraindication to administration of tacrolimus (Prograf or Advagraf), or other macrolides.
* Subject is unlikely to comply with the visits scheduled in the protocol or has a history of non-compliance.
* Subject has evidence of active liver disease or the presence of a chronic active hepatitis B or C within 1 month prior to kidney transplant surgery.
* Recipient or donor is seropositive for human immunodeficiency virus.
* Subject has active systemic infection requiring the use of antimicrobial agents within 1 week prior to kidney transplant surgery.
* Subject has current malignancy or a history of malignancy (within the past 5 years), except non- metastatic basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix that has been treated successfully.
* Subject has medical or psychological conditions which would preclude compliance with the study requirements.
* Subject has any condition, including any uncontrolled disease state other than end-stage kidney disease, that constitutes an inappropriate risk or a contraindication for participation in the study, or that could interfere with the study objectives, conduction, or evaluation.
* Female subject who breastfeed or donate ova starting at screening and throughout the study period.
* Male subject who donate sperm starting at screening and throughout the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed graft function (DGF) | Up to Day 7 after transplantation
  DGF is defined as dialysis requirement during the first post-transplant week (7 days).

SECONDARY OUTCOMES:
Incidence of acute rejection (AR) | Up to Month 6 after transplantation
  The reporting of AR includes any biopsy-proven or clinically-suspected rejection of a subject after transplantation.
Renal function assessed by estimated glomerular filtration rate (eGFR) | Up to Month 6 after transplantation
  eGFR will be derived using the abbreviated Modification of Diet in Renal Disease (MDRD) formula.
Renal function assessed by serum creatinine | Up to Month 6 after transplantation
  Serum creatinine will be measured from serum sample collected.
Renal function assessed by urea nitrogen | Up to Month 6 after transplantation
  Urea nitrogen will be measured from serum sample collected.
Subject survival | Up to Month 6 after transplantation
  Subject survival is the time from the date of transplantation to the date of death or the date of the last follow-up. Subject survival will be estimated using Kaplan Meier estimates and compared by log rank test.
Graft survival | Up to Month 6 after transplantation
  Graft survival is an estimate of the probability of the transplant functioning at a finite time after transplantation. Graft survival will be calculated from the date of transplantation to the date of irreversible graft failure or the date of the last follow-up during the period when the transplant is still functioning or to the date of death.
Safety assessed by incidence of treatment-emergent adverse events (TEAEs) | Up to Month 7 after transplantation
  Adverse events (AEs) will be coded using the latest version of MedDRA. TEAE is defined as any AE following the transplantation until the end of the study.
Safety assessed by incidence of serious adverse events (SAEs) | Up to Month 7 after transplantation
  AE is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Number of participants with laboratory test abnormalities and/or AEs | Up to Month 7 after transplantation
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Month 7 after transplantation
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead electrocardiograms (ECG) abnormalities and/or AEs | Up to Month 7 after transplantation
  ECG will be performed in the supine position after the subject has been breathing quietly for 5 minutes. Any clinically significant adverse changes on the ECG will be reported as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma China, Inc.
Locations (14):
- China (14):
  - Site CN08608, Beijing
  - Site CN08619, Beijing
  - Site CN08609, Changsha
  - Site CN08604, Guangzhou
  - Site CN08614, Hangzhou
  - Site CN08617, Hangzhou
  - Site CN08610, Nanjing
  - Site CN08618, Nanjing
  - Site CN08612, Shanghai
  - Site CN08603, Tianjin
  - Site CN08621, Wenzhou
  - Site CN08602, Wuhan
  - Site CN08613, Wuhan
  - Site CN08605, Xi'an

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Oliveras L, Lopez-Vargas P, Melilli E, Codina S, Royuela A, Coloma Lopez A, Fava A, Manonelles A, Couceiro C, Lloberas N, Cruzado JM, Montero N. Delayed initiation or reduced initial dose of calcineurin-inhibitors for kidney transplant recipients at high risk of delayed graft function. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD014855. doi: 10.1002/14651858.CD014855.pub2. PMID 40197799
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — http://www.trialsummaries.com/Study/StudyDetails?id=14639&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — http://www.clinicaltrials.astellas.com/study/506-MA-3186/